CLINICAL TRIAL: NCT03501199
Title: Comparison of Different Materials Contribution to Immediate Implants Stability With Resonance Frequency Analysis
Brief Title: Comparison of Different Materials Contribution to Implants Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gökhan Gürses, Research Assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NecmettinEU-Dentistry
Record Dates: First submitted 2018-03-23; First posted 2018-04-18 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-12

CONDITIONS: Dental Implant Failure Nos
Keywords: immediate implant placement
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRF Group (Experimental): PRF is will be used in immediate dental implant placement.
  Interventions: Other: platelet-rich fibrin placement; Procedure: tooth extraction; Procedure: immediate implant placement; Other: collagen membran placement; Procedure: raising flap
- Graft Group (Experimental): The xenogenic graft is will be used in immediate dental implant placement.
  Interventions: Other: xenogenic graft placement; Procedure: tooth extraction; Procedure: immediate implant placement; Other: collagen membran placement; Procedure: raising flap
- Control Group (Experimental): No extra material is will be used in immediate dental implant placement.
  Interventions: Other: no extra material; Procedure: tooth extraction; Procedure: immediate implant placement; Other: collagen membran placement; Procedure: raising flap

INTERVENTIONS:
Other: platelet-rich fibrin placement — filling the buccal gap with platelet-rich fibrin after immediate dental implant placement
  Arms: PRF Group
Other: xenogenic graft placement — filling the buccal gap with xenogenic graft after immediate dental implant placement
  Arms: Graft Group
Other: no extra material — filling the buccal gap with no material after immediate dental implant placement
  Arms: Control Group
Procedure: tooth extraction — extraction of tooth which is unrestorable
Procedure: immediate implant placement — putting dental implant into a socket which has been prepared with compatible drills
Other: collagen membran placement — placing collagen membran on extraction socket after dental implant placement to cover all
Procedure: raising flap — raising the buccal flap with two vertical incision to cover extraction socket for primary closure

SUMMARY:
The investigators will use two types of material(PRF-Xenograft) in the buccal gap after immediate dental implant placement. The study design has three groups PRF, graft, and control group. The patients will randomly be assigned to groups by envelop method. The resonance frequency analysis device(Osstell) will be used to measure primary and secondary stabilization. Then the investigators will evaluate each materials' contribution to stability.

Pre-op and 9th month Post-op CBCTs will evaluate about bone loss in mesial-distal and horizontal dimensions.

ELIGIBILITY:
Inclusion Criteria:

* medically healthy,
* only one maxillary aesthetic region(incisors or premolars) tooth which has two adjacent teeth is indicated for extraction.
* intact buccal socket walls
* the gap between buccal socket wall to implant sholder at least 2 mm.

Exclusion Criteria:

* relevant tooth has more than one root,
* smoking,
* alcohol abuse,
* pregnancy,
* immune-suppressive patients,
* any systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Primer Stabilization-Resonance Frequency Analysis | at 0 day
  initial measurement after placement by Osstell device

SECONDARY OUTCOMES:
Seconder Stabilization-Resonance Frequency Analysis | 120th day
  secondary measurement after placement by Osstell device
Mesial-Distal and Horizontal Bone Loss | 9th month
  The alveolar bone loss between first day to 9th month

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Esen, Study Chair — Consultant; Gökhan Gürses, Study Director — Care Provider
Locations (1):
- Necmettin Erbakan University, Faculty of dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No